CLINICAL TRIAL: NCT05386654
Title: AI/ML Algorithm Training and Validation for the imPulse™ Tor System Self-Directed Systolic & Diastolic Blood Pressure Monitor.
Brief Title: imPulse™ Tor System Self-Directed Cuffless Blood Pressure Monitoring
Status: Completed | Type: Observational
Sponsor: Level 42 AI, Inc. (Industry)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: L42CVP-0005
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: AI-driven, Self-directed Blood Pressure Monitoring
Keywords: infrasound; vibroacoustic; capacitive ECG; electric potential sensor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: imPulse™ Tor System — Self-directed blood pressure data capture
  Other Names: Clinical reference gold standard sphygmomanometer

SUMMARY:
Self-measured, non-invasive accurate blood pressure monitoring continues to be a major challenge for automated vital sign measurement systems. The general notion is that with reliable, self-administered BP monitoring in the clinic and at home, health care providers will be able to diagnose hypertension among individuals at an early stage, including high risk patients in the community, and more quickly assess if prescribed treatment plans are working. The imPulse™ Tor System detects 1) audible and inaudible low-frequency, low-amplitude sounds generated by the body, including arterial pulse waveforms, and 2) ECG-derived heart cycle identification, which can be combined with the vibroacoustic data to estimate blood pressure. The imPulse™ Tor has undergone preliminary testing. In this pilot study, we collect data from health care workers for algorithm training and validation study to achieve medical grade device AAMI/ISO and IEEE standards compliance.

DETAILED DESCRIPTION:
Hypertension (HTN) is a major risk factor for cerebrovascular morbidity and mortality, yet its identification can be delayed due to lack of overt symptoms, relying on Blood Pressure (BP) measurements for diagnosis. Several BP monitoring techniques are used in clinics and hospitals, and there is also an outpatient method that is used for 24-hour BP monitoring, based on a sphygmomanometer. The general notion is that with frequent, reliable, self-directed BP monitoring in the clinic and at home, health care providers will be able to diagnose hypertension among individuals at an early stage, including high-risk patients in the community, and more quickly assess if prescribed treatment plans are working. However, non-invasive self-administered blood pressure monitoring continues to be a major challenge for automated vital sign measurement systems.

To circumvent the limitations of current systems of interval hemodynamic measurement and increasing demands on healthcare providers, a non-invasive automated self- directed vital sign monitor that can integrate into hospital early warning systems and warn healthcare providers of deteriorating vital sign parameters would be of significant value. This study aims to provide proof of concept for a portable device that measures vital signs (blood pressure, heart rate, and blood oxygen saturation) using biophysical pneumatics and hydraulics, vibroacoustics, and multi-lead ECG that aims to produce results that are as good as a sphygmomanometer-based device and pulse oximeter, without the need for a circumferential pressure device/sphygmomanometer on the arm.

ELIGIBILITY:
Inclusion Criteria:

• Participants are limited to clinical staff and first-responders who work at the UC Davis C Street Clinics in the Sports and Spine suites.

Exclusion Criteria:

* History of major neck surgeries
* Unable to sit and stand upright comfortably for 2 minutes
* Unable to obtain or has contraindication to upper extremity blood pressure reading
* Unable to perform self-measurements using the imPulse™ Tor device
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteer healthcare worker cohort
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
imPulse™ Tor System Blood Pressure Prediction | bid/1week
  Following AI/ML algorithm training and validation the difference between predicted systolic, diastolic, and mean arterial pressure predictions of the imPulse™ Tor and gold-standard measurement of an electronic blood pressure cuff will be less than 2.5 mmHg in at least 90% of the measurements, less than 5 mmHg in at least 92.5% of the measurements and less than 10 mmHg in at least 95% of the measurements.

SECONDARY OUTCOMES:
imPulse™ Tor Heart Rate Prediction | bid/1week
  Following AI/ML algorithm training and validation, there is no significant difference (p-values >0.05) in the comparisons of electronic blood pressure cuff pulse measurement and imPulse™ Tor estimations for HR measurements (BPM).
imPulse™ Tor Oxygen Saturation Prediction | bid/1week
  Following AI/ML algorithm training and validation, the imPulse™ Tor can predict oxygen saturation (a proposed fifth vital sign) with an overall classification accuracy > 85% for the SpO2 class "< 84%", "85 to 91%" and "> 92%", respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- UCD Sports Medicine, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
Pilot study data for algorithm training using different AI/ML approaches.